CLINICAL TRIAL: NCT00273065
Title: Phase 1 Study of Local Infiltration of Neosaxitoxin as a Local Anesthetic
Brief Title: Local Anesthetic Properties of Neosaxitoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chile (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HCUCH-AR-NEOSAX-0001
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2007-02

CONDITIONS: Healthy Volunteers
Keywords: Local Anesthetic; Neosaxitoxin
MeSH Terms: interventions — neosaxitoxin

INTERVENTIONS:
Drug: Neosaxitoxin

SUMMARY:
The purpose of this study is to evaluate the local anesthetic properties of neosaxitoxin in humans

DETAILED DESCRIPTION:
Neosaxitoxin is a phycotoxins that reversible block the voltage-gated sodium channels at neuronal level. Its activity is express as blocking the axonal conduction, stopping the propagation of the nerve impulse. The objective of the present work is to evaluate the neosaxitoxin efficacy and safety as local anesthetic in a human trial

Methods: Randomized, double-blind, placebo-controlled trial, with 10 healthy volunteers. The anesthetic effect will be evaluated using a standardized human sensory and pain model. TSA Neurosensory analyser and Von Frey Technique will be used to evaluate five parameters: sensory threshold for warm and cold, pain thresholds for heat and cold and mechanical touch perception threshold.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males with the abilities to understand and respond the tests to perform

Exclusion Criteria:

* Use of any oral analgesics at least ten days before the study
* Drugs abuse history
* Showing at the clinical examination any signal of psychiatric disorder

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2005-05; Study Completion 2005-09

PRIMARY OUTCOMES:
Neural blockade of five parameters:
sensory threshold for warm
sensory threshold for cold
pain thresholds for heat
pain thresholds for cold
mechanical touch perception threshold
Measurements at 1,3,6,9,12,16,24 and 48 hrs after the injections

SECONDARY OUTCOMES:
Pain on injection (VAS Score 0-10)
Blood sample at 1 hour
Orine sample at 4 hours after the injection, in order to determine amounts of neosaxitoxin

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Rodriguez-Navarro, MD, Principal Investigator — University of Chile; Nestor Lagos, PhD, Principal Investigator — Faculty of Medicine, University of Chile
Locations (1):
- Henry Mayer Center, Hospital Clínico Universidad de Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Result] Rodriguez-Navarro AJ, Lagos N, Lagos M, Braghetto I, Csendes A, Hamilton J, Figueroa C, Truan D, Garcia C, Rojas A, Iglesias V, Brunet L, Alvarez F. Neosaxitoxin as a local anesthetic: preliminary observations from a first human trial. Anesthesiology. 2007 Feb;106(2):339-45. doi: 10.1097/00000542-200702000-00023. PMID 17264729